CLINICAL TRIAL: NCT02311738
Title: The Effect of Exercise and Genes on Energy Expenditure, Appetite and Quality of Life in Morbidly Obese Patients
Brief Title: Exercise and Genes in Obese (EGO)
Acronym: EGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jarle Berge (Other)
Collaborators: University of South-Eastern Norway (Other); Vestfold University College (Other); Duke University (Other); University of Agder (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Jarle Berge, PhD-Fellow, Sykehuset i Vestfold HF
Organization: Sykehuset i Vestfold HF (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EGO
Record Dates: First submitted 2014-06-26; First posted 2014-12-08 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: Exercise and Genes in Obese (EGO)
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High intensity training group (Experimental): HIE will consist of the following:
  1. 10 minute warm up at 70% of maximal heart rate.
  2. 4 minute exercise intervals at 90-95% of maximal heart rate.
  3. 4 minute interval bouts repeated 4 times.
  4. Between each bouts there will be a 3 minute active recovery at 70% of maximal heart rate
  5. After all four bouts are completed; 5 minute cool-down at 70% of maximal heart rate.
  Interventions: Other: Training intensity intervention
- Moderate intensity training group (Experimental): MIE will consist of the following:
  1. 10 minute warm up at 50% of maximal heart rate.
  2. 35 minutes exercise at 70% of maximal heart rate.
  3. 4 minute cool-down at 50% of maximal heart rate.
  Interventions: Other: Training intensity intervention

INTERVENTIONS:
Other: Training intensity intervention — High intensity training group describes the group performing high intensity exercise intervention. Moderate intensity training group describes the the group performing moderate exercise intervention
  Other Names: EGO-HIT

SUMMARY:
Regular exercise has several positive health effects including increased physical fitness and muscle mass. It is well known that increased muscle mass is associated with increased resting energy expenditure which may facilitate weight loss and maintenance. Previous studies have, however, failed to show any consistent association between the intensity of physical exercise and energy expenditure, or relate the variance in these adaptations to genetic variability. Whether high-intensity exercise (HIE) is associated with improved health related quality of life in severely obese patients remains unknown.

This PhD-project is based on a planned randomised controlled study including 50 or more treatment seeking morbidly obese patients who will be randomised to either a 24 week moderate-intensity exercise (MIE) programme or a 24 week high-intensity exercise (HIE) programme. The investigators main hypothesis is that patients randomised to the HIE-program will achieve higher energy expenditure during rest and physical activity after treatment than those allocated to the MIE-programme. In addition, the investigators hypothesise that the HIE-group will achieve a better health related quality of life than the MIE-group after treatment. The investigators also hypothesize that inter-individual variability in adaptation to the two training regimens may be due to genetic factors. If the investigators hypotheses are confirmed, this project might have beneficial clinical implications for future obesity treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Treatment seeking weight stable morbidly obese patients (BMI ≥ 40 kg/m2 or BMI 35 to 39.9 kg/m2 with ≥ 1 co morbidity) attending the outpatient Obesity Center, Vestfold Hospital Trust, will be informed about this RCT .

Exclusion Criteria:

* Uncompensated heart failure
* Recent myocardial infarction or stroke (<½ years)
* Severe arrhythmia or heart failure
* Unstable angina pectoris
* Renal failure
* Pregnancy
* Severe eating disorders
* Active substance abuse
* Being on a diet
* Taking medication known to affect appetite or metabolism (including thyroxin).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure during physical activity | 0, 8, 12 and 24 weeks
  Energy expenditure (EE) during volitional activity will be measured with ergo-spirometry tests one week before the exercise intervention period starts, and repeated after each exercise period. Increasing the aerobic work capacity is supposed to give the same proportional increase in energy expenditure at any given maximal intensity.

SECONDARY OUTCOMES:
Resting metabolic rate | 0, 8, 12 and 24 weeks
  Resting metabolic rate will be measured with ergo-spirometry test one week before the exercise intervention period starts, and repeated after each exercise period. Increasing the aerobic work capacity is supposed to give increased resting metabolic rate.
Cardiorespiratory fitness | 0, 8, 12 and 24 weeks
  Exercise may have a positive effect on cardiorespiratory fitness and will be measured with ergo-spirometry test
Body mass index | 0, 8, 12 and 24 weeks
  Exercise may have a positive effect on weight change and will be calculated as weight in kilograms divided by height in meters squared
Waist circumference | 0, 8, 12 and 24 weeks
  Exercise may have a positive effect on waist circumference and will be measured midway between the bottom edge of the lower rib and upper iliac crest in the horizontal plane.
Fat mass and fat free mass | 0, 8, 12 and 24 weeks
  Exercise may have a positive effect on body composition and will be measured with the bioelectrical impedance analyser Tanita BC-418
Appetite control | 0,12 and 24 weeks
  Patient self-appraisal of hunger and fullness will be assessed during fasting and after a standardised breakfast every 30 minutes (for a period of 3hours) using visual analogue scales.
Genetic susceptibility | 0, 8, 12 and 24 weeks
  We hypothesize that inter-individual variability in adaptation/response to the two training regimens may also be due to genetic factors. We have designed a gene panel consisting of recognized and previously reported risk genes/variants with flanking sequences relevant for exercise (VO2max), participation in physical activity, obesity, diabetes, asthma and obesity related sub-phenotypes. The panel covers 1.2 Mb and includes 299 genes (exons with exon-intron junctions) and 1468 intronic and intergenic SNPs. Next-generation sequencing will be performed using a gene panel of selected genes/genetic regions by Illumina Nextera technology. The method involves enzymatic fragmentation of DNA and probe-based enrichment. The samples will be sequenced (paired-end, 2x100 bp) on a HiScanSQ. All wet lab methods (with other gene panels) are ISO15189 certified and in routine use at Unit for Medical Genetics at Telemark Hospital.
Short form health survey (RAND-36) | 0,12 and 24 weeks
  RAND-36 is a 36-item measure of generic HRQOL consisting of eight additive subscales (Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health) and two summary scores each based on four subscales (Physical Component Summary and Mental Component Summary). Scores on all subscales range from 0 to 100. Summary-scores will be norm-based, with mean (SD) 50 (10). Higher scores on all scales represent better HRQOL.
Impact on Weight Questionnaire (IWQOL-Lite) | 0,12 and 24 weeks
  IWQOL-Lite is a 36-item measure of generic HRQOL consisting of eight additive subscales (Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health) and two summary scores each based on four subscales (Physical Component Summary and Mental Component Summary). Scores on all subscales range from 0 to 100. Summary-scores will be norm-based, with mean (SD) 50 (10). Higher scores on all scales represent better HRQOL.
Weight-Related Symptom Measure (WRSM) | 0,12 and 24 weeks
  WRSM is a 20-item measure for the presence and distress of 20 weight-related symptoms. The distress scores of the symptoms are reported on a six-point likert scale. Two summary scores are calculated; an additive score of presence of symptoms ranging from 1 to 20 and a symptom distress score for all symptoms. Symptom distress scores range from 0 to 100, with higher scores indicating a higher or worse total symptom distress.
Power of Food scale (PFS) | 0,12 and 24 weeks
  PFS assess both the psychological impact and respondent's responsiveness to a food-abundant environment. This is a 15-item scale whose items pertain to three situations: food being readily available in the environment but not physically present, food is physically present, but not tasted, and food is first tasted but not already consumed. The three subscales is scored 0-100 with higher scores indicating greater eating problems.
Binge Eating Scale (BES) | 0,12 and 24 weeks
  BES comprise 16 items assessing binge eating problems. Additive scores range between 0-46, with higher scores indicating greater problems. Cut-off scores have been established to determine binge severity, with "severe" represented by scores > 27, "moderate" by scores 18-26, and "mild-none" by scores < 17.
Three Factor Eating Questionnaire (TFEQ -R21) | 0,12 and 24 weeks
  TFEQ -R21 is a 21-item questionnaire covering eating behavior domains: the cognitive restraint scale (6 items) assesses control over food intake and influence over body weight and body shape; the emotional eating scale (6 items) measures the propensity to overeat in relation to negative mood states, e.g., when feeling lonely, anxious, or depressed; and, the uncontrolled eating scale (9 items) assesses the tendency to lose control over eating when feeling hungry or when exposed to external stimuli
Body weight change | 0, 8, 12 and 24 weeks
  Exercise may have a positive effect on weight change

OTHER OUTCOMES:
Substrate oxidation | 0, 8, 12 and 24 weeks
  Exercise may have a positive effect on substrate oxidation (for example fat oxidation) and will be measured with ergo-spirometry tests
Hip circumference | 0, 8, 12 and 24 weeks
  Exercise may have a positive effect on hip circumference and will be measured on the widest part of the hip in the horizontal plane.
Daily activity | 0, 17 and 24 weeks
  Exercise can affect daily activity. Measurements of 24-hour activity during free living will be performed with accelerometer (ActiGraph wGT3x-BT, Pensacola, FL, USA). The 24-hour activity expressed as daily activity counts per minute (Vector magnitude, CPM). The registrations will last for 24 hours during 7 days including the weekend.
Total energy intake | 0 and 24 weeks
  Exercise can affect total energy intake. A 180 items food frequency questionnaire developed in Norway and validated to assess habitual diet among men and women, was will be used. The dietary data will be entered by scanning, using the teleform program (10.0) (Datascan, Oslo, Norway). Daily intake of foods, energy and nutrients will be calculated using software (KBS version 7.3 2017; developed at the institute of Basic Medical Sciences, University of Oslo). The software is based on Norwegian food composition table (Norwegian Food Composition Database 2017. Norwegian Food Safety Authority)

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, professor, Study Director — The Hospital of Vestfold
Locations (6):
- Duke University School of Medicine, Durham, North Carolina, United States
- Norway (5):
  - Vestfold University College, Horten, Raveien
  - Telemark University College, Bø
  - University in Agder, Kristiansand
  - Norges Teknisk-naturvitenskapelig Universitet, Trondheim
  - Vestfold Hospital Trust, Tønsberg

REFERENCES:
- [Derived] Berge J, Hjelmesaeth J, Kolotkin RL, Storen O, Bratland-Sanda S, Hertel JK, Gjevestad E, Smastuen MC, Helgerud J, Bernklev T. Effect of aerobic exercise intensity on health-related quality of life in severe obesity: a randomized controlled trial. Health Qual Life Outcomes. 2022 Feb 24;20(1):34. doi: 10.1186/s12955-022-01940-y. PMID 35209911
- [Derived] Berge J, Hjelmesaeth J, Hertel JK, Gjevestad E, Smastuen MC, Johnson LK, Martins C, Andersen E, Helgerud J, Storen O. Effect of Aerobic Exercise Intensity on Energy Expenditure and Weight Loss in Severe Obesity-A Randomized Controlled Trial. Obesity (Silver Spring). 2021 Feb;29(2):359-369. doi: 10.1002/oby.23078. PMID 33491314